CLINICAL TRIAL: NCT03798717
Title: The Effect of Acute, Passive Heating on Glucose Tolerance in Individuals With Type 2 Diabetes Mellitus: a Randomised, Balanced Crossover, Control Trial
Brief Title: To Bathe or Not to Bathe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Ant Shepherd, Senior Lecturer, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 003AS
Record Dates: First submitted 2018-12-20; First posted 2019-01-10 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will lie in a semi recumbent position in minimal clothing for the entirety of the visit. Initially, participants will be cannulated and blood samples drawn.every 30 min of each experimental visit. Following cannulation an 180 min OGTT (75g) will commence in a thermoneutral room (~ 23C). During the OGTT, HR will be measured continuously, whilst blood pressure, deep body temperature (rectal probe) and resting metabolic rate will be assessed every 30 min.
- Pre OGTT (Experimental): Condition 2 will employ identical procedures to condition 1, except thirty minutes into the OGTT, the participant will be immersed into an immersion tank (~39oC) for 60 min. Water temperature will be manipulated as required to achieve and maintain a target Trec at 38.5 oC using water between 37.5 and 39oC, and then participants will be removed horizontally back into the thermoneutral room for the reminder of the OGTT. Participants will be towel dried and given a towelled robe to wear.
  Interventions: Diagnostic Test: Heating
- Post OGTT (Experimental): Condition 3 will employ identical procedures to condition 2, with the exception that the heating via immersion will start as soon as the participant is instrumented (and following a 15 min rest period) and the OGTT will commence 30 min after the 60 min immersion time for a further 180 min.
  Interventions: Diagnostic Test: Heating

INTERVENTIONS:
Diagnostic Test: Heating — Warm water immersion
  Other Names: Bath
  Arms: Post OGTT; Pre OGTT

SUMMARY:
Type 2 diabetes mellitus (T2DM) is characterised by chronic high blood sugar concentration (hyperglycaemia) and insulin resistance leading to a reduction in insulin sensitivity. These hyperglycaemic excursions can seriously impact metabolic, micro and macrovascular health. The total cost of the direct and indirect care of individuals with diabetes (~90% T2DM) in the UK (United Kingdom) is £23.7 billion, equating to ~20% of the annual national health service (NHS) budget, with this projected to become unsustainable. Low-cost interventions to improve glycaemic control in these individuals are therefore warranted. Current interventions include pharmaceuticals, exercise and calorie restrictive diets. Pharmaceutical interventions carry a high financial cost, while exercise and diet programmes have a low adherence rate in individuals with T2DM.

Heat therapy offers one potential low cost therapy. Immersion in a hot tub for 30 mins.day-1 for 10 days has been shown to reduce fasting plasma [glucose] and HbA1c in individuals with T2DM, which may be explained by acute (e.g. muscle) and chronic (e.g. reduced inflammatory status and increased heat shock proteins (HSP)) adaptations, although experimental evidence for these hypothesis are sparse. Other potential benefits include improved glycaemic control, insulin sensitivity, elevated resting metabolic rate and improved micro- and macrovascular function.

The aim of the present study is to determine whether acute hot water immersion can improve glucose tolerance in individuals with T2DM and whether it is more beneficial to undertake this before or after a OGTT (oral glucose tolerance test).

DETAILED DESCRIPTION:
Visit 1 (consent, screening and familiarisation) During visit 1, participants will give their informed consent, followed by a health screening questionnaire. In addition to the health screening questionnaire, medical history and a blood sample will be collected and analysed for a full blood count, glycated haemoglobin (HbA1c), liver and kidney function. Finally, a resting electrocardiogram (ECG) will also be recorded and then examined for irregularities, where a clinical decision will be made on further participation to the study by consultants at QA (Queen Alexandra) hospital. Participants will then be shown the rest of the equipment and taken through the procedure for the next 3 visits and, if the participant is happy to continue the study, the next visit will be organised.

Visit 2, 3 and 4 Participants will arrive at the laboratory at ~9 am for conditions 1 and 2 and 8 am for condition 3. Prior to a 15 min resting period (supine) before any measures are taken participants will be asked to insert a rectal thermistor (participants will be given clear instructions using the investigator's SoPs (standard operating procedure)). Condition 1, 2 and 3 will be balanced and participants randomly allocated to begin the study in either visit 2, 3 or 4 using a blinded member of the team.

For all visits (see figure 2), participants will lie in a semi recumbent position in minimal clothing (bathing shorts and a t-shirt) for the entirety of the visit. Initially, participants will be cannulated (Versatus winged and ported IV cannula, Terumo, Japan) and blood samples drawn for analysis of osmolality (Lithium Heparin (LH) tubes BD (Becton, Dickinson and Company), USA) plasma [glucose] (Fluoride/Oxalate tubes, BD, USA), [insulin] (Ethylenediaminetetraacetic acid (EDTA) K2, BD, USA), and [eHSP70 (extracellular heat shock protein 70)] (EDTA K2, BD, USA) at baseline and every 30 min of each experimental visit. Following cannulation an 180 min OGTT (75g) (Rapilose OGTT solution, Penlan healthcare, Japan) will commence in a thermoneutral room (~ 23oC). A maximum of 18 mL of blood being drawn at each time point (max 126 mL per visit). To maintain the patency of the cannula and to reduce the risk of infection, after every sample is taken, 5 mL of saline will be flushed through the cannula. Then before every sample is taken, 2.5 mL of blood will be drawn out of the cannula to ensure any remaining saline will not interfere with the samples and data interpretation (additional 17.5mL per visit). During the OGTT, HR (heart rate) (via electrocardiogram) will be measured continuously, whilst blood pressure (M5-1, Omron, Japan), deep body temperature (rectal probe) and resting metabolic rate (indirect calorimetry) (Quark CPET (cardiopulmonary exercise test), Cosmed, Italy) will be assessed every 30 min.

Condition 2 will employ identical procedures to condition 1, except thirty minutes into the OGTT, the participant will be immersed into an immersion tank (~39oC) for 60 min. Water temperature will be manipulated as required to achieve and maintain a target Trec at 38.5 oC using water between 37.5 and 39oC, and then participants will be removed horizontally back into the thermoneutral room for the reminder of the OGTT. Participants will be towel dried and given a towelled robe to wear. Condition 3 will employ identical procedures to condition 2, with the exception that the heating via immersion will start as soon as the participant is instrumented (and following a 15 min rest period) and the OGTT will commence 30 min after the 60 min immersion time for a further 180 min (see figure 2 for a schematic).

ELIGIBILITY:
The participants must meet all of the following criteria to be considered eligible for the study:

* Male or female (either post-menopausal or in the early-follicular phase (3-5 days after the onset of menstruation) of the menstrual cycle), aged 35 years or above.
* Diagnosed with T2DM as defined by the WHO (World Health Organisation).
* Participant is willing and able to give informed consent for participation in the study.
* Participant is able to understand and fully cooperate with the study protocol.

Exclusion Criteria

The participant may not enter / be withdrawn from the study if any of the following apply:

* Severe peripheral neuropathy (to the point to which they cannot sense temperature)
* Uncontrolled hypertension (≥180 systolic / 100 diastolic mmHg)
* Taking any medication which may interfere with data interpretation or safety
* Who have had a myocardial infarction or cerebro-vascular event
* Any cardiac abnormalities which restrict hard exercise
* Current smokers or who have stopped within 3 months
* Participant is unable to understand and/or fully cooperate with the study protocol
* Any other serious medical condition which would interfere with data interpretation or safety will be excluded from participation.
* Any skin conditions including ulcerations

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to release IPD (individual patient data), until all avenues of further funding have been exhausted.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 440 individuals were screened for eligibility (200 clinical letters, 40 from day events and 200 from local diabetes education group). 420 declined and 0 were excluded. Once participants were randomly allocated to arm sequence 5 withdrew before starting. Three in-between experimental visits. Twelve completed the study and data analysed.
Pre-assignment Details: Participants were excluded from the study before assignment to groups if they did not pass screening criteria. Balanced randomisation of order in which individuals completed each arm (cross-over) was carried out. Therefore there was an equal number of individuals completing all combinations of arms.
Groups:
- Control - Pre OGTT - Post OGTT: Participants first underwent a 3 h OGTT (oral glucose tolerance test) with no passive heating. Then approximately a week later underwent a 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT. Then, approximately a week underwent a 1 h bout of passive heating 30 min into a 3 h OGTT.
- Control - Post OGTT - Pre OGTT: Participants first underwent a 3 h OGTT with no passive heating. Then, approximately a week underwent a 1 h bout of passive heating 30 min into a 3 h OGTT. Then approximately a week later underwent a 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT.
- Pre OGTT - Control - Post OGTT: Participants first underwent a 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT. Then, approximately a week later underwent a 3 h OGTT with no passive heating. Then, approximately a week underwent a 1 h bout of passive heating 30 min into a 3 h OGTT.
- Pre OGTT - Post OGTT - Control: Participants first underwent a 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT. Then, approximately a week underwent a 1 h bout of passive heating 30 min into a 3 h OGTT. Then, approximately a week later underwent a 3 h OGTT with no passive heating.
- Post OGTT - Control - Pre OGTT: Participants first underwent underwent a 1 h bout of passive heating 30 min into a 3 h OGTT. Then, approximately a week later underwent a 3 h OGTT with no passive heating. Then, approximately a week later underwent 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT.
- Post OGTT - Pre OGTT - Control: Participants first underwent underwent a 1 h bout of passive heating 30 min into a 3 h OGTT. Then, approximately a week later underwent 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT. Then, approximately a week later underwent a 3 h OGTT with no passive heating.
Period: Overall Study
Arm/Group | Control - Pre OGTT - Post OGTT | Control - Post OGTT - Pre OGTT | Pre OGTT - Control - Post OGTT | Pre OGTT - Post OGTT - Control | Post OGTT - Control - Pre OGTT | Post OGTT - Pre OGTT - Control
Started | 4 | 3 | 3 | 4 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 2 | 1 | 1 | 2 | 1 | 1
Not completed — Failed Screening | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — COVID-19 (coronavirus disease) Lockdown | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Individuals with T2DM
Groups:
- Control - Pre OGTT - Post OGTT: Participants first underwent a 3 h OGTT with no passive heating. Then approximately a week later underwent a 1 h bout of passive heating ending 30 min before undertaking a 3 h OGTT. Then, approximately a week underwent a 1 h bout of passive heating 30 min into a 3 h OGTT.
- Total: Total of all reporting groups
Arm/Group | Control - Pre OGTT - Post OGTT | Control - Post OGTT - Pre OGTT | Pre OGTT - Control - Post OGTT | Pre OGTT - Post OGTT - Control | Post OGTT - Control - Pre OGTT | Post OGTT - Pre OGTT - Control | Total
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 3 | 3 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 2 | 1 | 2 | 9
  >=65 years | 2 | 2 | 2 | 2 | 2 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 0 | 1 | 5
  Male | 3 | 2 | 2 | 3 | 3 | 2 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean AUC (Area Under the Curve) Plasma [Glucose]
Description: Does an acute bout of passive, warm water therapy reduce plasma [glucose]? Units for AUC are AU (arbitrary units) which have been derived from the trapezoidal method and have been published as such. Trapezoidal method: AUC = Δx ((y0/2)+y1+y2+y3+...+(yn/2)).
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: Individuals with T2DM (type 2 diabetes mellitus)
Measure: Mean (Standard Deviation); unit: AU
Groups:
- Control: Participants will lie in a semi recumbent position in minimal clothing for the entirety of the visit. Initially, participants will be cannulated and blood samples drawn every 30 min of each experimental visit. Following cannulation an 180 min OGTT (75g) will commence in a thermoneutral room (~ 23C). During the OGTT, HR (heart rate) will be measured continuously, whilst blood pressure, deep body temperature (rectal probe) and resting metabolic rate will be assessed every 30 min.
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 12 | 12 | 12
AU | 1677 (386) | 1797 (340) | 1662 (364)

2. Secondary Outcome: Change in Plasma [Insulin]
Description: Does plasma [insulin] reduce more if the passive, warm water therapy is conducted before or after the OGTT?
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: Individuals with T2DM
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 12 | 12 | 12
µU/mL | 75.18 (68.94) | 48.79 (35.11) | 79.86 (63.91)

3. Secondary Outcome: Mean Insulin Sensitivity
Description: Does insulin sensitivity increase following an acute bout of warm water therapy? Calculation of insulin sensitivity is measured in AU which have been derived from the Gutt method and have been published as such. Gutt insulin sensitivity = [75,000 + (G0-G120) × 0.19 × BW]/(120 × log [(I0 + I120)/2] × [(G0 + G120)/2]). Where G = plasma [glucose], I = plasma [insulin] and BW = body weight.
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: Individuals with T2DM
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 12 | 12 | 12
AU | 52.00 (11.56) | 47.45 (13.86) | 56.51 (13.85)

4. Secondary Outcome: Change in Fuel Utilisation
Description: Does carbohydrate and fat (RER) utilisation alter during and following an acute bout of warm water therapy?
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: Individuals with T2DM
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 12 | 12 | 12
kcal | 263 (33) | 278 (40) | 304 (38)

5. Secondary Outcome: Change in Cardiovascular Status
Description: Does heart rate (variability) change during or after an acute bout of warm water therapy?
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: 0 participants analysed due to immersion for passive heating causing too much noise in the data for it to be valid.
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in eHSP70 (Extracellular Heat Shock Protein 70)
Description: Does eHSP increases during and following an acute bout of warm water therapy?
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: Individuals with T2DM
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 8 | 8 | 8
pg/mL | 324 (154) | 507 (112) | 364 (81)

7. Secondary Outcome: Change in Inflammatory Status
Description: Does inflammatory status (IL-6 & IL-10) change during or after an acute bout of warm water therapy?
Time Frame: Visit 2, 3 and 4. 3 times in total, until study completion, approximately 8 weeks
Population: 0 participants analysed due to lack of funds as a result of the COVID-19 pandemic. Data for this has not been collected and will not be in the future.
Arm/Group | Control | Pre OGTT | Post OGTT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3h for the OGTT plus the 1 h of passive heating in the passive heating arms at Visit 2, 3 and 4. 3 times in total, until study completion, up to approximately 8 weeks.
Description: Safety population included all participants who underwent the OGTT and passive heating.
Arm/Group | Control | Pre OGTT | Post OGTT
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=12) | Pre OGTT (N=12) | Post OGTT (N=12)
Pain on cannulation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Participant experienced pain on cannulation
Vasovagal syncope (Investigations) | 0 (0) | 0 (0) | 2 (2) — Vasovagal syncope (1 on existing the water, 1 during study assessments).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT03798717/Prot_SAP_000.pdf